CLINICAL TRIAL: NCT01333176
Title: Community-based Screening for Diabetes Using a Validated Point-of-care HbA1c Assay in a British Columbia First Nations Community
Brief Title: Point of Care HbA1c as a Screening Test for Type 2 Diabetes in First Nations
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Vancouver General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H10-02551
Record Dates: First submitted 2011-04-05; First posted 2011-04-11 (Estimated); Last update posted 2012-04-25 (Estimated); Status verified 2012-04

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Hb A1c screening for diabetes in aboriginals
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All volunteers have HbA1c test (Experimental): All candidates receive same procedure
  Interventions: Procedure: Point-of-care "finger-poke" HbA1c determination.; Procedure: HbA1c blood test; Procedure: HbA1c finger poke test; Procedure: Blood test

INTERVENTIONS:
Procedure: Point-of-care "finger-poke" HbA1c determination. — All volunteers receive finger-poke HbA1c test. Result: If < 6: Offered a requisition to have gold standard testing for diabetes screening. If 6-6.5: Given requisition for FBG, HbA1c and OGTT. If A1c result >6.5: Counseled that they may have diabetes. Given requisition as above.
  Estimates about how many have undiagnosed diabetes will be calculated.
  1. Did the clients who were counseled to do so get follow-up blood tests?
  2. Were all the formal diagnostic tests performed?
  3. Did the formal tests correlate to the POC HbA1c test or was there significant discrepancy? Thus is this new test for diagnosing diabetes confirmed as a valid test for screening in First Nation Communities in Canada?
  4. Did the family physicians find this useful?
  Other Names: Ames/Bayer DCA 2000 Hemoglobin A1c Assay
Procedure: HbA1c blood test — All candidates will have a HbA1c blood test (Finger poke)
Procedure: HbA1c finger poke test — All study candidates will have the same HbA1c test performed
Procedure: Blood test — HbA1c blood test
Procedure: Blood test — HbA1c finger poke blood test

SUMMARY:
1. Purpose

   * to estimate the prevalence of undiagnosed diabetes mellitus and pre-diabetes in a BC First Nation community
   * to determine the utility of community based screening by examining how many positively screened people follow up with the recommended subsequent testing and family physician visit
   * to determine if point-of-care HbA1c test (Ames/Bayer DCA 2000) correlates with the confirmatory fasting and 2 hour post challenge blood glucose tests.
2. Hypothesis The Point-of-Care test will correlate well with the gold standard diagnostic tests and prove to be a useful tool for community-based screening. This test obviates the need for fasting and repeat glucose tolerance testing.

DETAILED DESCRIPTION:
This is a screening for prevalence study.

The Seabird Island Band's health department serves a large catchment area of approximately 3000 First Nation members. The team of physicians, nurses, and technicians will invite communities to participate in diabetes screening events. In conjunction with the community health workers, we will be facilitating diabetes awareness in the community through the provision of large scale screening Two types of events will be held. An initial "Open House" event and a second event in the form of an afternoon "Diabetes Awareness" event later in the year.

With the assistance of community leaders and the Seabird Island Health Unit staff, we will utilize materials such as posters and flyers available from the Health unit both to increase awareness of diabetes and to advise of the awareness/screening events. For the Community Event there will be a community dinner served at the end of the afternoon for all who attended.

Community members of Seabird Island will be invited for screening through posters hung in gathering spaces and high traffic areas. Notices will be put in the community newsletter.

They will be given information about the screening study and will give informed consent by way of a formal consent form. If younger than 18, consent will be obtained from parents or guardians. Identity will be concealed by using study numbers for individuals; a master list linking names and PHNs to the study numbers will be kept by the Seabird Island lead for the study at Seabird Island in a locked cabinet in a locked office. Primary and Co-investigators will receive only anonymized data. This is the wish of the community and is in keeping with OCAP principles.

Tests and Procedure:

Point of care (finger poke) HbA1c using Ames/Bayer DCA 2000 POC analyzer system will be used for screening.

1. If the A1c test result is < 6%: Will be offered to have a fasting and 2 hour after glucose drink test (OGTT) the next day. Otherwise will be counseled to follow up in one year with their Primary Care Physician or attend another screening opportunity
2. If A1c result is 6-6.5: Given lab requisition for fasting blood sugar and HbA1c and 2 hour after glucose drink test (OGTT). Advised to get follow up blood work tomorrow (in some cases this will be available in the community) and advised to see their family physician. If the family physician is not a Seabird physician, a letter will be sent to the physician informing him of the screening event and the screening results. Counseled about health promotion and diabetes and meaning of A1c result.
3. If A1c result is >6.5: Counseled that they may have diabetes. Given requisition to obtain a fasting and two hour post glucose drink test (OGTT) tomorrow and advised to see their family physician. Counseled about health promotion and diabetes and meaning of A1c result.

If history of gestational diabetes and not retested - given requisition for 75 g OGTT and counseled to follow up with family physician. If the family physician is not a Seabird physician, a letter will be sent to the physician informing him of the screening event and the screening results. Counseled about health promotion and diabetes and meaning of A1c result.

If blood pressure > 140/90 - counseled to follow up with family physician. If the family physician is not a Seabird physician, a letter will be sent to the physician informing him of the screening event and the screening results.

The Seabird lead will be notified of the blood results and record them along with the screening results. Anonymized data will be forwarded to the investigative team. We recognize that a small proportion of the sample (approximately 15%) that have non-Seabird physicians may not have follow-up data available.

All participants will have received information regarding diet, lifestyle, and diabetes prevention. They will also be given general counseling regarding the role of balance in health, and the fact that the traditional medicine wheel identifies Physical, Spiritual, Mental and Emotional aspects of health that affect blood glucose levels.

Estimates will be made (based on this sample of the population) about how many people have undiagnosed diabetes in this community, that is the number not known to have self-reported diabetes but who have an A1c test >6.5%. Specifically, if the A1c test is greater than 6.5% this is considered diagnostic of diabetes (by current American Diabetes Association standards) This will be compared to the number who have diabetes based on a fasting glucose > 7 mmol/L and/or 2 hour post glucose drink blood glucose test > 11 mmol/L on follow up testing (by current Canadian Diabetes Association guidelines) As well, comparison of the reverse will be made, namely those with elevated fasting and/or post glucose drink values but who had normal A1c values (<6.5%)

Additional outcomes:

1. Did the clients who were counseled to do so actually obtain the follow-up blood tests? (Historically, such patients often decline to obtain the tests requested).
2. Were all the follow-up blood tests performed? How many declined one or more of these tests, specifically the 2 hour post glucose drink test which is often refused).
3. Did the formal tests correlate to the POC HbA1c test or was there significant discrepancy? Thus is this test for diagnosing diabetes confirmed as a valid test for screening in First Nation Communities in Canada?
4. By one month post screening survey, how what percentage of family physicians found this useful?

Follow up information will be obtained and analyzed:

1. Dr. Fox (main Seabird physician) will be contacted 1 month after the screening day to follow up on patient visits and on outpatient blood work for which clients were given requisitions. He will be asked if he noticed any benefits of this program.
2. After 3 months, Dr. Fox will be re-contacted to check for outstanding results.
3. At 4 months, if follow-up blood work has not been performed, clients will be contacted individually by telephone by Seabird Health to be reminded and to find out why they did not follow through with the blood tests.

6) Statistical Analysis

Primary end point: How many clients (all of whom claimed not to have known diabetes) had HbA1c > 6.5%? This number indicates the prevalence of unknown diabetes in this First Nation community. And how many clients had a fasting glucose >7% and 2 hour post glucose drink glucose level >11%? Comparison of these two groups of results will indicate the correlation of the A1c test with the conventional glucose diagnostic tests in this First Nation population.

Secondary end points:

How many clients had an HbA1c > 6% but <6.5% and therefore have pre-diabetes. How many clients have hypertension with Blood pressure > 140/90. How many clients with a history of gestational diabetes and no follow up OGTT had diabetes (HbA1c >6.5%)

Sample size: If n=320 and we observe a prevalence of diabetes of 10%, then the absolute margin of error (the 95% confidence interval for the observed proportion) is +/- 3.3%, 19 times out of 20.

ELIGIBILITY:
Inclusion Criteria:

* Members of Seabird Island or surrounding communities
* self-identified as First Nation1
* 14 years old and older

Exclusion Criteria:

* Known diabetes
* age less than fourteen years old
* pregnancy or less than six weeks post-partum
* medications known to interfere with glucose metabolism
* acute illness,
* life-expectancy of less than six months

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Does the HbA1c identify the same individuals as fasting and 2-hr pc glucose tests to identify diabetes and pre-diabetes in a First Nation community | One Month between individual comparative samples; One year for recruitment of all subjects.
  We will obtain A1c, fasting glucose, and 2 hour post glucose drink glucose tests in First Nation volunteers. An A1c result of 6-6.4% will be considered diagnostic of pre-diabetes, a result ≥6.5% diabetes, a fasting glucose of 6.1-6.9 mmol/L pre-diabetes, and a fasting glucose ≥7 mmol/L, diabetes. Individual A1c results will be compared to fasting and 2 hour post glucose drink results. We will determine the sensitivity and specificity of the A1c test compared to the fasting and post glucose drink glucose tests.

SECONDARY OUTCOMES:
Provide estimates of prevalence of diabetes and prediabetes in a First Nation community | One year
  To estimate the prevalence of undiagnosed diabetes mellitus and pre-diabetes in a random sample of the population from Seabird Island First Nation community.
To identify the response rate of "gold standard" diabetes testing in a First nation community | One Year
  To determine what percentage of those screened "positive" or "at risk" follow up with recommendations for formalized testing and follow up with family physician.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica MacKenzie-Feder, MD, Study Director — University of British Columbia; Sandra Sirrs, MD, Study Director — Universithy of British Columbia
Locations (1):
- Vancouver General Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Piette JD, Milton EC, Aiello AE, Mendoza-Avelares MO, Herman WH. Comparison of three methods for diabetes screening in a rural clinic in Honduras. Rev Panam Salud Publica. 2010 Jul;28(1):49-57. doi: 10.1590/s1020-49892010000700008. PMID 20857021